CLINICAL TRIAL: NCT02299466
Title: Home Total Parenteral Nutrition (HTPN) in Canada: A New Website Based Patient Registry
Brief Title: Registry for Patients Receiving Intravenous Nutrition at Home
Acronym: HTPN
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Nutrition Society (Other); Baxter Healthcare Corporation (Industry); Ontario Medical Supply (Unknown)
Responsible Party: Principal Investigator, Johane Allard, MD, FRCPC, University Health Network, Toronto
Other Study IDs: 03-0845-AE
Record Dates: First submitted 2014-10-24; First posted 2014-11-24 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Parenteral Nutrition, Home
Keywords: parenteral nutrition; complications; indications; long-term administration; HTPN
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of study is to build a Canadian HTPN Registry to collect pertinent demographic and clinical data on the HTPN population in Canada and to determine the factors affecting survival, complications and TPN-dependency. These results will help establish standards of practice and develop future multi-center studies. This will greatly benefit the HTPN patient population.

DETAILED DESCRIPTION:
The HTPN Registry is website based. Only users inside of Canada will be able to access the website. All data is held in Ontario, Canada and is governed by Ontario and Canadian privacy and security laws. The entry point into the registry will be through a website www.htpnregistry.ca, using a specific HTPN program password for data entry. A code and date of birth will be used to identify each patient. Patient data will be kept confidential and be entered by a member of the TPN team from each participating program. Participating programs will have access to their own database and will be able to compare their patient population to the one of the entire registry. Data entered into the registry will include: 1) Patient demography 2) Nutritional assessment 3) Medications 4) Indications for HTPN 5) Gastrointestinal anatomy following surgeries 6) HTPN regimen 7) Current blood work 8) Vascular access 9) Hospitalizations 10) Survival, 11) Liver complications 12) Metabolic bone disease 13) quality of life. In addition, information regarding each HTPN program will be captured: organization of the TPN team, number of patients under the program, diagnosis and reasons for HTPN, source of funding, geographical coverage, home care utilization, providers. Data will be entered every two years by the one or more HTPN staff monitoring the patients. The data can be entered directly into the website or case report forms can be used to collect the data from the patient charts and facilitate data input into the website.

All patients will be followed prospectively until discontinuation of TPN or death. Descriptive statistics will be performed.

For the entire HTPN population, probability of survival, chronic cholestasis, complicated home parenteral nutrition related liver disease, line infection and metabolic bone disease will be calculated using the Kaplan-Meier method. As of February 2014, 433 patients (85 from UHN) have been entered into the Canadian HTPN registry. The recruitment and data collection is expected to continue for at least 5 more years (until 2019). Participating HTPN programs are: Toronto (Toronto General Hospital, St. Michael's Hospital), Hamilton (Hamilton Health Sciences),Winnipeg (St. Boniface General Hospital), Edmonton (Capital Health/University Of Alberta), Calgary (Foothills Medical Centre), British Columbia (BC Home Parenteral Nutrition Program) and Montreal (McGill University).

ELIGIBILITY:
Inclusion Criteria:

* Patients with long-term administration of home total parenteral nutrition Age >18 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving home total parenteral nutrition (HTPN)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2005-12 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | bi-annually up to 10 years, discontinuation of HTPN or death
  Body weight, body mass index

SECONDARY OUTCOMES:
Patient characteristics | baseline
  Age, sex, medical history
Medications | bi-annually up to 10 years, discontinuation of HTPN or death
  Immunosuppressors, motility agents, antidiarrheal, sedatives, antidepressors, anticoagulants, insulin, inhibitors of acid secretion, medication to treat liver disease (eg. urso, carnitine, choline…), medication to treat metabolic bone disease (eg. iv/oral calcium, vitamin D, biphosphonate, calcitonin,… are collected from the charts
Indications for HTPN | bi-annually up to 10 years, discontinuation of HTPN or death
  Short bowel, motility disorder, cancer, surgical complications, pancreatic disorders, other causes of malabsorption
Gastrointestinal anatomy | bi-annually up to 10 years, discontinuation of HTPN or death
  Anatomy as described in medical records
HTPN regimen | bi-annually up to 10 years, discontinuation of HTPN or death
  Energy, amino acids, lipids, fluid, electrolytes, vitamins, trace elements
Current blood work | bi-annually up to 10 years, discontinuation of HTPN or death
  Complete blood count , biochemistry including liver enzymes, total protein, albumin, prealbumin, vit B12, red blood cell folate, iron studies,international normalized ratio /prothrombin time /partial thromboplastin time , cholesterol, triglycerides, trace elements;parathyroid hormone , 24-hr urine oxalate
Vascular access | bi-annually up to 10 years, discontinuation of HTPN or death
  type of catheter, number of lumens, changes in vascular access, complications (line sepsis, occlusion)
Hospitalizations | bi-annually up to 10 years, discontinuation of HTPN or death
  Number/year and TPN related or not TPN related
Survival | bi-annually up to 10 years, discontinuation of HTPN or death
  Alive, death: causes, TPN-related or not TPN-related
Liver complications | bi-annually up to 10 years, discontinuation of HTPN or death
  Diagnosis, abdominal ultrasound results, liver biopsy results
Metabolic Bone Disease | bi-annually up to 10 years, discontinuation of HTPN or death
  Bone mineral density results, fracture risk and reported fractures
Quality of life based on Karnofsky performance scale | bi-annually up to 10 years, discontinuation of HTPN or death
  Karnofsky performance scale (0-100 point scale)

CONTACTS AND LOCATIONS:
Overall Officials: Johane Allard, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (10):
- Canada (10):
  - Foothills Medical Centre, Calgary, Alberta
  - Captial Health/University Of Alberta, Edmonton, Alberta
  - BC Home Parenteral Nutrition Program, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Hopital St-Luc, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - Saskatchewan Adult HTPN Program, Regina, Saskatchewan

REFERENCES:
- [Result] Saqui O, Fernandes G, Allard JP. Quality of life analysis during transition from stationary to portable infusion pump in home parenteral nutrition patients: a Canadian experience. Nutr Clin Pract. 2014 Feb;29(1):131-41. doi: 10.1177/0884533613516129. Epub 2013 Dec 17. PMID 24347531
- [Result] Abdalian R, Fernandes G, Duerksen D, Jeejeebhoy KN, Whittaker S, Gramlich L, Allard JP. Prescription of trace elements in adults on home parenteral nutrition: current practice based on the Canadian Home Parenteral Nutrition Registry. JPEN J Parenter Enteral Nutr. 2013 May-Jun;37(3):410-5. doi: 10.1177/0148607112463074. Epub 2012 Oct 12. PMID 23064256
- [Result] Abdalian R, Saqui O, Fernandes G, Allard JP. Effects of manganese from a commercial multi-trace element supplement in a population sample of Canadian patients on long-term parenteral nutrition. JPEN J Parenter Enteral Nutr. 2013 Jul;37(4):538-43. doi: 10.1177/0148607112454543. Epub 2012 Jul 24. PMID 22829428
- [Result] Jawa H, Fernandes G, Saqui O, Allard JP. Home parenteral nutrition in patients with systemic sclerosis: a retrospective review of 12 cases. J Rheumatol. 2012 May;39(5):1004-7. doi: 10.3899/jrheum.110896. Epub 2012 Mar 1. PMID 22382342
- [Result] Fernandes G, Kaila B, Jeejeebhoy KN, Gramlich L, Armstrong D, Allard JP. Canadian home parenteral nutrition (HPN) registry: validation and patient outcomes. JPEN J Parenter Enteral Nutr. 2012 Jul;36(4):407-14. doi: 10.1177/0148607111434599. Epub 2012 Feb 10. PMID 22326909
- [Result] Aljarallah B, Fernandes G, Jeejeebhoy KN, Gramlich LM, Whittaker JS, Armstrong D, Duerksen DR, Allard JP. The Canadian Home Total Parenteral Nutrition (HTPN) Registry: vitamin K supplementation and bone mineral density. JPEN J Parenter Enteral Nutr. 2012 Jul;36(4):415-20. doi: 10.1177/0148607111431983. Epub 2012 Feb 1. PMID 22301331
- [Result] Raman M, Gramlich L, Whittaker S, Allard JP. Canadian home total parenteral nutrition registry: preliminary data on the patient population. Can J Gastroenterol. 2007 Oct;21(10):643-8. doi: 10.1155/2007/217897. PMID 17948134
- [Derived] Clermont-Dejean NM, Schwenger KJP, Salazar E, Colombo FF, Lu Z, Lou W, Gramlich L, Whittaker S, Armstrong D, Jurewitsch B, Raman M, Duerksen DR, McHattie JD, Murthy S, Allard JP. Home parenteral nutrition patients on mixed oil lipid emulsion have a higher rate of hospitalizations compare to those on soybean oil- a prospective 2-year cohort study. Clin Nutr. 2021 Jul;40(7):4616-4623. doi: 10.1016/j.clnu.2021.06.012. Epub 2021 Jun 17. PMID 34229267